CLINICAL TRIAL: NCT06336512
Title: Trimester Sequential Estimation of Serum Zonulin Overrides Glucose Homeostasis Biomarkers for Prediction of Gestational Diabetes Mellitus
Brief Title: Trimester Sequential Estimation of Serum Zonulin as a Predictor of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed K Zaineldin, Lecturer of Obstetrics & Gynecology, Faculty of Medicine, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC.28.1.2024
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Newly Pregnant Women with singleton fetus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- serum zonulin (Other)
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Estimation of Zonulin by ELISA from the Blood samples which were obtained at time of pregnancy .

SUMMARY:
Gestational diabetes mellitus (GDM) is the development of glucose intolerance (GI) during pregnancy in a previously normoglycemic (NG) woman and associated with insulin resistance (IR). GDM is the most prevalent metabolic disorder during pregnancy and became a major public health problem for being usually diagnosed and detected after 24 gestational weeks (GW), while its complications can occur much earlier and this may explain its burden on maternal and fetal welfare. Human zonulin is a surrogate marker of intestinal permeability and can be utilized as biomarker for intestinal barrier function. Zonulin-mediated increase in intestinal permeability plays a role in the pathogenesis of insulin resistance, obesity, DM and metabolic syndrome. The increasing global prevalence of GDM with its associated risk of poor pregnancy and long-term risks for the mother and the offspring may lead to the production of new generation of diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women with singleton fetus

Exclusion Criteria:

* Women with morbid obesity with body mass index ≥35 kg/m2;
* Had manifest DM, irrespective of being controlled or not;
* Bowel-related disorders;
* Autoimmune disorders;
* History of previous GDM.

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Estimation of Gestational DM | 8 months
  Relation between Serum Zonulin levels and Gestational Diabetes Mellitus

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El- Qalyobia, Egypt